CLINICAL TRIAL: NCT05489419
Title: Evaluation of Prehabilitation as a Strategy to Minimize Surgical Risk in Pancreatic Surgery: Efficacy and Determining Factors.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HCB/2020/0477
Record Dates: First submitted 2022-07-04; First posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-07

CONDITIONS: Pancreatic Neoplasms; Anesthesia
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prehabilitation (Experimental): Patients undergo prehabilitation during 3-4 weeks before undergoing pancreatic surgery.
  Interventions: Behavioral: Multimodal Prehabilitation

INTERVENTIONS:
Behavioral: Multimodal Prehabilitation — Physical and cardiopulmonary training, personalized nutrition and treatment of anxiety and depression.

SUMMARY:
Several studies in major abdominal surgery demonstrated that preoperative optimization of surgical patients through prehabilitation is associated with fewer postoperative complications. However, patients' response to preoperative optimization is unpredictable, and there are no studies confirming the real benefit in pancreatic surgery.

Aims: To assess the benefits of pre-rehabilitation in pancreatic surgery, and identify those factors associated with an effective optimization. Secondary aims: impact of prehabilitation on nutritional status, sarcopenia, quality of life, inflammation markers, postoperative complications and hospital stay compared to low-risk patients.

Design: An objective multimodal assessment will be performed on those patients who are candidates to pancreaticoduodenectomy (PD) to identify patients at high-risk of postoperative complications. These patients will undergo prehabilitation and response will be evaluated. Intervention:Multimodal Prehabilitation will include:

1. Physical and cardiopulmonary training followed by a personalized program according to basal aerobic capacity, patient circumstances and compliance, community-based and remote-controlled with information and communication technology (ICT).
2. Personalized nutrition program adapted to the underlying disease (exocrine insufficiency, cachexia and sarcopenia, diabetes).
3. Treatment of anxiety and depression.

Subjects: 56 consecutive patients who are high-risk candidates (anaerobic threshold 11ml/kg/min at CPET) for PD recruited at Hospital Clinic of Barcelona. Postoperative variables will be compared to low-risk patients evaluated during the same study period.

Analysis:

The main variable will be aerobic capacity (VO2max, AT). Secondary variables (before and after the program) will be nutritional status, sarcopenia, quality of life, inflammation markers and immune response, hospital stay, complications, 90-days mortality and costs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients eligible for pancreatic surgery (PD) who are considered high risk based on the findings of the CPET (anaerobic threshold, AU <11ml/kg/min) (Older P et al. Crit Care. 2004;8:369-72) and accepted as candidates for said surgery by the multidisciplinary committee of our Institution.

Exclusion Criteria:

* Non-elective surgery;
* Palliative surgery;
* Unstable respiratory or cardiac disease;
* Locomotor or cognitive limitations that prevent adherence to the program;
* Refusal to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of a multimodal prehabilitation | 4 weeks
  To evaluate the efficacy of a multimodal prehabilitation program in high risk surgical patients undergoing oncological resection of the pancreas in terms of improvement in aerobic capacity (peak oxygen consumption, anaerobic threshold) measured through a CPET.

SECONDARY OUTCOMES:
Evaluation of the adherence to the program | 30 days
  Assess the % of sessions that the patient has completed
Evaluation of sarcopenia after prehabilitation | 4 weeks
  Sarcopenia analyzed objectively with a CT scan.
Evaluation of the impact on perceived quality of life | 4 weeks
  Evaluation of the impact of the program in patient quality of life according EuroQol (Qual Life Res. 1999 ;8:303-10)
Evaluation of the impact on the inflammatory response after the intervention | 30 days
  Presence or abscence of Systemic Inflammatory Response Syndrome (SIRS) during the preoperative period. SIRS defined by two of the following criteria: Body temperature over 38 or under 36 degrees Celsius.
  Heart rate greater than 90 beats/minute Respiratory rate greater than 20 breaths/minute or partial pressure of CO2 less than 32 mmHg Leucocyte count greater than 12000 or less than 4000 /microliters or over 10% immature forms or bands.
Evaluation of the impact on the incidence of postoperative complications | 30 days
  Incidence of complications
Evaluation of complications severity | 30 days
  Complications according Clavien-Dindo Classification

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No